CLINICAL TRIAL: NCT07184424
Title: A Real-world Study on the Addition of Lenalidomide to Reverse Resistance After First-line Treatment Lenvatinib Combined With PD-1 Therapy in Advanced Hepatocellular Carcinoma
Brief Title: Real-world Study of Lenalidomide After First-line Treatment Lenvatinib With PD-1 in Advanced HCC
Acronym: Lenalidomide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dream-004
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: Lenalidomide; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): In clinical practice, for patients with hepatocellular carcinoma (HCC) who have received targeted therapy combined with immune checkpoint inhibitors as first-line treatment and subsequently experienced disease progression, lenalidomide capsules are incorporated into the regimen (administered orally on days 1-21, followed by a 7-day treatment-free interval, repeating every 28 days per cycle).
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — For patients with hepatocellular carcinoma who have experienced disease progression after receiving standard clinical treatment with lenvatinib in combination with PD-1 inhibitors, the addition of lenalidomide capsules to the three-drug combination therapy was followed by a 2-month follow-up liver imaging examination to observe changes in the target lesion and whether new lesions had developed in other areas.
  Other Names: lenalidomide capsules

SUMMARY:
This study is a real-world, single-arm, observational study primarily collecting data on patients with hepatocellular carcinoma who experienced disease progression after receiving lenvatinib in combination with PD-1 inhibitors as part of routine clinical practice, and evaluating the efficacy of adding lenalidomide to their treatment regimen.

DETAILED DESCRIPTION:
This study is a real-world, single-arm, observational study primarily collecting data on patients with hepatocellular carcinoma who experienced disease progression after receiving lenvatinib in combination with PD-1 inhibitors as part of routine clinical practice, and evaluating the efficacy of adding lenalidomide to their treatment regimen.

The treatment drugs used in this study are: Lenvatinib mesylate capsules (imported or domestically produced), immunotherapy: PD-1 inhibitors (approved for marketing in China and abroad), and Lenalidomide capsules.

The study population was divided into three groups: 1. Patients with advanced, unresectable hepatocellular carcinoma treated with lenvatinib in combination with a PD-1 inhibitor, who showed imaging evidence of disease progression (defined as an increase in the maximum diameter of the primary tumor by more than 20% or the emergence of new lesions) and were planned to receive additional treatment with lenalidomide; 2. Patients currently receiving lenvatinib plus PD-1 inhibitor plus lenalidomide therapy due to disease progression; 3. Patients who have previously received lenvatinib plus PD-1 inhibitor plus lenalidomide therapy; Participants in categories 1 and 2 will sign an informed consent form and be enrolled in this study for symptomatic treatment. Category 3 study participants, who have previously received this treatment regimen, cannot obtain informed consent. Therefore, this study has applied for informed consent waiver for Category 3 study participants (this option is not available in the reporting system).

According to standard clinical treatment principles, collect hematological examination data from patients one week and one month after receiving combination therapy with lenvatinib + PD-1 inhibitor + lenalidomide.Collect hematological and imaging examination data two months after combination therapy, and evaluate the imaging data at the two-month mark to determine whether the tumor has progressed.Each observation cycle lasts two months.

Enrollment standard：

1.Age ≥ 18 years old 2.Patients with hepatocellular carcinoma who previously received lenvatinib and PD-1 inhibitors and whose tumors progressed on imaging (enhanced MRI, enhanced CT, or PET-CT) were treated with lenalidomide.

3.Expected survival period exceeding 3 months 4.Patients with a history of other malignant tumors who have been disease-free for more than 2 years after initial treatment (such as non-melanoma skin cancer or cervical carcinoma in situ) 5.Participants of childbearing age agreed to use contraception during the study period Exclusion standard：

1. Fibrous plate layer or sarcomatous HCC or mixed type HCC-ICC
2. Currently participating in and receiving other experimental treatments, or participating in an immune checkpoint inhibitor study and receiving study treatment.
3. Previously underwent solid organ transplantation, diagnosed with immunodeficiency
4. Bleeding from esophageal or gastric varices within 3 months prior to enrollment
5. Hepatic encephalopathy in the past 6 months, or obvious ascites at the time of enrollment.
6. Active infection requiring systemic treatment
7. CTCAE grading Platelet count < 50 × 10⁹/L or neutrophil count < 1 × 10⁹/L
8. Pregnant or breastfeeding women
9. Patients with myocardial ischemia or myocardial infarction classified as grade II or higher according to the Common Terminology Criteria for Adverse Events (CTCAE), uncontrolled arrhythmia
10. Patients who have previously used pomalidomide or thalidomide
11. Patients who have previously received CTLA-4 in combination with PD-1/PD-L1 inhibitors
12. Other situations deemed unsuitable for participation in this trial by researchers

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Patients with hepatocellular carcinoma who previously received lenvatinib and PD-1 inhibitors and whose tumors progressed on imaging (enhanced MRI, enhanced CT, or PET-CT) were treated with lenalidomide；
* Expected survival period exceeding 3 months;
* Patients with a history of other malignant tumors who have been disease-free for more than 2 years after initial treatment (such as non-melanoma skin cancer or cervical carcinoma in situ);
* Participants of childbearing age agreed to use contraception during the study period;

Exclusion Criteria:

* Fibrous plate layer or sarcomatoid HCC or mixed type HCC-ICC;
* Currently participating in and receiving other experimental treatments;
* Previously underwent solid organ transplantation, diagnosed with immunodeficiency;
* Bleeding from esophageal or gastric varices within 3 months prior to enrollment;
* Hepatic encephalopathy in the past 6 months, or obvious ascites at enrollment;
* Active infection requiring systemic treatment;
* CTCAE grading Platelet count < 50 × 10⁹/L or neutrophil count < 1 × 10⁹/L
* Pregnant or breastfeeding women;
* Patients with myocardial ischemia or myocardial infarction graded CTCAE grade II or higher, or uncontrolled arrhythmia;
* Patients who have previously used pomalidomide or thalidomide;
* Patients who have previously received CTLA-4 in combination with PD-1/PD-L1 inhibitors;
* Other situations deemed unsuitable for participation in this trial by researchers;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
1 year PFS | Following the administration of lenalidomide combination therapy, imaging examinations of lesion sites should be performed every two months to assess tumor status.
  The time from enrollment in the clinical study until the first evidence of disease progression or death.Every two month, up to 1 year
OS | For one year or longer, until death
  From the start of treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: GONG LI, phD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No